CLINICAL TRIAL: NCT01910584
Title: Prospective Study of the Influence on Quality of Life and Sexual Function of the Novasure Endometrial Ablation in the Treatment of Menorrhagia
Brief Title: Quality of Life and Sexual Function of the Novasure Endometrial Ablation in Menorrhagia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shu-Qin Chen (Other)
Responsible Party: Sponsor-Investigator, Shu-Qin Chen, associate professor of gynaecology and obstetrics, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: First-GYN-SYSU-2012
Record Dates: First submitted 2013-07-20; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2012-09

CONDITIONS: Quality of Life; Sexual Activity
Keywords: quality of life; sexual activity; Novasure endometrial ablation; menorrhagia
MeSH Terms: conditions — Sexual Behavior; Menorrhagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Novasure treated group: patients diagnosed menorrhea were treated with novasure endometrial ablation
  Interventions: Procedure: Novasure endometrial ablation

INTERVENTIONS:
Procedure: Novasure endometrial ablation — Novasure endometrial ablation is the second generation endometrial ablation treatment aimed to cure the dysfunctional uterine bleeding(DUB),including menorrhagia.

SUMMARY:
The aim of this study is to investigate the influence on the quality of life and sexual function before, 6 month and one year after Novasure Endometrial Ablation in the treatment of Menorrhagia.

DETAILED DESCRIPTION:
patients diagnosed menorrhagia scheduled for Novasure Endometrial Ablation because of menorrhagia between november, 2012 and november, 2014 are enrolled to this study.

patients are asked to complete preoperative questionnaires considering Health Related Quality of Life questionnaire(HRQoL) and sexual Female Sexual Functioning Index questionnaire(FSFI). Same questionnaires will also be completed six months and one year after operation.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of menorrhagia
* family complete
* normal endometrial pathology
* had not been referred specifically for surgery
* with normal uterine cavity

Exclusion Criteria:

* pregnancy or demand to preserve fertility
* acute reproductive tract inflammation or urinary tract inflammation
* pathology demonstrate endometrial cancer or precancerous change
* acute pelvic inflammation
* intrauterine device(IUD) in uterus
* depth of uterine cavity less than 4cm or more than 10cm
* pathologic myometrium( such as history of Hysteromyomectomy or classical cesarean section)

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients diagnosed menorrhagia scheduled for Novasure endometrial ablation in The First Affiliated Hospital between November 2012 and November 2015
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life and Sexual Function before, six month and one year after the Novasure Endometrial Ablation | one year after Novasure Endometrial Ablation
  Quality of life assessed with Health Related Quality of Life questionnaire(HRQoL) before, six month and one year after the Novasure Endometrial Ablation; Sexual Function measured with Female Sexual Functioning Index questionnaire(FSFI) before, six month and one year after the Novasure Endometrial Ablation

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Zhong Yao, PhD & MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun yat-sen University, Guangzhou, Guangdong, China